CLINICAL TRIAL: NCT00152711
Title: Impact of nCPAP Treatment on Liver Function in Patients With Sleep Apnea Syndrome and Nonalcoholic Steatohepatitis: A Prospective Cross Over Trial
Brief Title: Impact of nCPAP Treatment on Liver Function in Patients With Sleep Apnea Syndrome and Nonalcoholic Steatohepatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PHRC 03-07
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2007-02-13 (Estimated); Status verified 2005-09

CONDITIONS: Sleep Apnea Syndrome; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Sleep Apnea Syndromes; Non-alcoholic Fatty Liver Disease

INTERVENTIONS:
Device: nCPAP

SUMMARY:
This study aims to evaluate the impact of nasal continuous positive airway pressure (nCPAP) treatment on liver enzymes in patients with sleep apnea syndrome and nonalcoholic steatohepatitis. Using a cross over design, the evolution of liver enzymes will be evaluated in 40 patients during a consecutive period of 6 weeks, with and without nCPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old
* Nonalcoholic steatohepatitis proven by liver biopsy
* Sleep apnea syndrome proven by polysomnography with an apnea-hypopnea index > 10 events/hour
* Informed consent

Exclusion Criteria:

* Psychiatric disorder
* Other cause of liver disease
* Professional driver

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Gagnadoux, Principal Investigator — UH Angers
Locations (1):
- University Hospital Angers, Angers, France